CLINICAL TRIAL: NCT01238068
Title: Comparison of the Results of Treatment by Gamma Nail Versus Dynamic Hip Screw for Unstable Intertrochanteric Hip Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: ortal segal, TASMC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TAMSC-10-OS-10-357-CTIL
Record Dates: First submitted 2010-10-26; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-10

CONDITIONS: Intertrochanteric Fractures of the Hip

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Gamma nail, fracture stabilization, better walking (Active Comparator)
  Interventions: Device: gamma nail stryker

INTERVENTIONS:
Device: gamma nail stryker — for acute unstable pertrochantric fractures the subjects will be treated randomaly with either Gamma nail device Vs Dynamic hip screw

SUMMARY:
The study hypothesis is the the results of the use of Gamma nail will be superior to the use of Dynamic hip screw for unstable intertrochantric hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* patients diagozied with acute intertrochantric unstable fracture
* a minimum minimental score of 6
* ability to walk 500 meters indepedently

Exclusion Criteria:

* pathological fracture
* multiple fractures
* neurological conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
hip function score | 1 year
  at the last clinical visit (1 year) the patient will perform hip score testing and record.

SECONDARY OUTCOMES:
x-ray, surgical outcome | 1 year
  in the last clincial visit x ray finding will be record and the overall surgical outcome (infection, bleeding etc.) will be record

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical center, Tel Aviv, Israel

REFERENCES:
- [Derived] Lewis SR, Macey R, Gill JR, Parker MJ, Griffin XL. Cephalomedullary nails versus extramedullary implants for extracapsular hip fractures in older adults. Cochrane Database Syst Rev. 2022 Jan 26;1(1):CD000093. doi: 10.1002/14651858.CD000093.pub6. PMID 35080771